CLINICAL TRIAL: NCT05478954
Title: Seasonal Malaria Chemoprevention in Burkina Faso : Chemoprevention Efficacy Study
Brief Title: Chemoprevention Efficacy Study in Burkina Faso
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Malaria Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SMCBFPHASE1
Record Dates: First submitted 2022-07-15; First posted 2022-07-28 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Malaria
Keywords: Seasonal-Malaria-Chemoprevention
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Intervention Model Description: Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sulfadoxine-Pyrimethamine + Amodiaquine (SPAQ) (Experimental): Children aged 3-59 months will receive SPAQ during the study period.
  Interventions: Drug: Sulfadoxine pyrimethamine; Drug: Amodiaquine

INTERVENTIONS:
Drug: Sulfadoxine pyrimethamine — Sulphadoxine is a slowly eliminated sulphonamide. It is used in a fixed dose combination of 20 parts sulphadoxine with 1 part pyrimethamine given orally or intramuscularly.
  The medicine is no longer recommended for the treatment of malaria. However, it is being used for Intermittent Preventive Treatment during pregnancy (IPTp) and as a co-packaged combination with amodiaquine for seasonal malaria chemoprevention.
  Sulphadoxine is readily absorbed from the GIT. It is widely distributed in body tissues and fluids and crosses the placenta into foetal circulation. It is also readily detectable in breast milk. It is excreted predominantly as the unchanged drug.
  Other Names: SP
Drug: Amodiaquine — Amodiaquine is a Mannich base 4 amino-quinoline that interferes with parasite haem detoxification. It is more effective than chloroquine in both chloroquine sensitive and resistant P. falciparum infections. However, there is cross-resistance between chloroquine and amodiaquine.
  It is readily absorbed in the GIT and rapidly converted in the liver to the active metabolite, desethylamodiaquine. Desethylamodiaquine is responsible for all the antimalarial effect. Adverse effect of amodiaquine includes abdominal discomfort and vomiting weakness and when used for prophylaxis it causes agranulocytosis. Amodiaquine is recommended as a partner drug in artemisinin based combination therapy.
  Other Names: AQ

SUMMARY:
The aim of this study is to determine whether Seasonal Malaria Chemoprevention (SMC) remains effective in the health district of Nanoro in the Centre-Ouest region or Boussé in the Plateau Central region. It also aims to assess the protective efficacy of the antimalarial drugs used in SMC in the target population and to investigate levels of parasite resistance in the study districts. According to the results, this trial should provide the evidence needed to change the drugs used in SMC.

A Type II hybrid effectiveness-implementation study design will be used to evaluate the effects of a clinical intervention on relevant outcomes whilst collecting information on implementation. It is designed to determine feasibility and effectiveness of an innovative intervention, as well as the protective efficacy of the antimalarial drugs used. The study consists of two components: 1) Conducting a prospective cohort study to determine the protective efficacy of the drug combination Sulfadoxine-Pyrimethamine and Amodiaquine (SPAQ) (if SPAQ provides 28 days of protection from infection) and whether drug concentrations and/or resistance influence the duration of protection; 2) Conducting a resistance markers study in symptomatic patients in the research district.

DETAILED DESCRIPTION:
This cohort study aims to evaluate the effects of a clinical intervention on relevant outcomes whilst collecting information on implementation.

The study uses pragmatic implementation research with the objective of contributing to the development of practical recommendations for health policy, practice and potential scale up. It is designed as an implementation study to determine effectiveness and protective efficacy to gather evidence of the potential impact on health outcomes. Five monthly cycles of SMC will be implemented between July and October 2022 in one district, Nanoro, in Centre Ouest region.

The study will comprise the following two components:

1. A prospective protective efficacy cohort study to determine if SPAQ provides 28 days of protection from infection and whether drug concentrations and/or resistance influence the duration of protection
2. A resistance markers study in children 3-59 months in the two research districts plus the two standard intervention districts to measure changes in resistance marker prevalence over time (pre and post within the same year and between years)

ELIGIBILITY:
Inclusion Criteria:

* Children between 3-59 months
* Being resident in the project area
* Afebrile with no other malaria associated symptoms in the past 48 hours or at time of recruitment
* Consent to participate in the study obtained
* Can comply with 3 day DOT of standard SPAQ regimen (day 0-2)
* Willingness and ability of the childs guardians to comply with the study protocol for the duration of the study including all dry blood spot and slide collections

Exclusion Criteria:

* Symptoms of malaria (tympanic fever ≥ 37.5 °C or history of fever in past 48 hours)
* Known allergy to medicine provided
* Receiving a sulfa-based medication for treatment or prophylaxis, including co-trimoxazole (trimethoprim-sulfamethoxazole).
* Individuals receiving azithromycin due to the antimalarial activity of azithromycin.
* Severe malnutrition according to WHO guidelines
* Recruited in cross sectional surveys or any other SMC studies.

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Chemoprevention failure as defined by qPCR positive parasites or malaria slide positive parasites | One month
  Malaria slides and dry blood spots (DBS) taken at days 0,7,14, 21, 28 of a one month drug administration cycle will be analysed to detect parasitemia in children treated with SPAQ. Chemoprevention failure has occured if a malaria slide is positive for parasites 7 days or more after drug administration or if a qPCR detects low level parasitemia at the end of the administration cycle (one month).
Prevalence of antimalarial resistance markers among chemoprevention failures (as defined in outcome 1) | One month
  All Dried blood spots (DBS) will be analysed for malaria mutation genotypes (dhfr, dhps, Pfcrt, pfmdr1) on baseline and endline and additionally throughout the cycle if a chemoprevention failure (as defined in outcome 1) has occured.
Drug concentrations of Sulfadoxine-pyrimethamine and amodiaquine among chemoprevention failures (as defined in outcome 1) | One month
  Drug concentrations of SPAQ will be analyzed on all samples (taken at days 7,14,21,28 throughout the one month cycle) in order to be linked to chemoprevention failures as defined in outcome 1.

SECONDARY OUTCOMES:
Prevalence over time of parasites with dhfr/dhps/pfcrt/pfmdr1 mutations in symptomatic children with a positive diagnostic test residing in districts where SMC is implemented | Five months
  The outcome measure to meet the secondary objective is the prevalence of molecular markers associated with SP (codons 108, 51 and 59 in dhfr and 437, 540 and 581 in dhps) and amodiaquine (codons 72-76 Pfcrt and 86, 184 and 1246 pfmdr1), as well as other markers of parasite genetic diversity, in blood samples collected from symptomatic children under five years with a positive RDT attending selected health facilities in areas with SMC.

CONTACTS AND LOCATIONS:
Overall Officials: Gauthier Tougri, Principal Investigator — NMCP Manager
Locations (1):
- Unité de Recherche Clinique de Nanoro, Nanoro, Burkina Faso

IPD SHARING:
Plan to Share IPD: No